CLINICAL TRIAL: NCT06430788
Title: Phase 2a/2b Study Emapalumab: A Window of Opportunity in Pediatric Aplastic Anemia
Brief Title: A Study of Emapalumab for Pediatric Aplastic Anemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23-278; FD-R-008175 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Aplastic Anemia; Cytopenia; Hypocellular Marrow
Keywords: pediatric aplastic anemia; aplastic anemia; cytopenia; hypocellular marrow; Emapalumab; Memorial Sloan Kettering Cancer Center; 23-278
MeSH Terms: conditions — Anemia, Aplastic; Cytopenia; Bone Marrow Failure Disorders | interventions — Emapalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Emapalumab, then Standard IST (Experimental): Participants will first receive Emapalumab for 6 weeks. After treatment with emapalumab, participants will receive standard IST with drugs called equine anti-thymocyte globulin (hATG) and cyclosporin (CsA) in addition to a lower dose of emapalumab
  Interventions: Biological: Emapalumab
- Emapalumab, then HCT (Experimental): Participants will first receive Emapalumab for 6 weeks. After treatment with emapalumab, participants will have a standard hematopoietic stem cell transplant (HCT).
  Interventions: Biological: Emapalumab

INTERVENTIONS:
Biological: Emapalumab — Emapalumab is an interferon gamma (IFNγ) blocking antibody
  Other Names: Gamifant

SUMMARY:
The purpose of this study is to find out whether upfront emapalumab treatment can help in sAA (Aplastic Anemia) treatment planning and increase the effectiveness of standard treatment options.

Funding Source- FDA OOPD

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing workup for suspected newly diagnosed sAA:

  * Patients with severe cytopenias and a hypocellular marrow concerning for sAA
  * Patients that meet the definition for suspected sAA (Camitta Criteria) as follows:

Marrow Cellularity: <25%, or 25-50% with <30% residual hematopoietic cells Peripheral cytopenias (at least 2 of 3) Absolute neutrophil count (ANC): <500 x 10^9/L Platelets: <20 x 10^9/L Absolute Reticulocyte Count: <60 x 10^9/L

* Patients that do not have evidence of leukemia or MDS
* Patients < 25 years of age at time of diagnosis
* Able to tolerate emapalumab and IST (with standard institutional organ function criteria)

Exclusion Criteria:

* Uncontrolled infection at presentation.
* Patients who have undergone previous treatment for sAA.
* Patients with known inherited bone marrow failure
* Patient who has completed a full workup for sAA including having results back from telomere testing, DEB and genetics (when applicable), as well as having an appropriate willing and available donor and would otherwise be admitted for HSCT within 2 weeks of enrolling on the trial
* Patients with leukemia or MDS
* Patient or parent or guardian unable to give informed consent or unable to comply with the treatment protocol including research tests.

Ages: 0 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2029-05-21 (Estimated); Study Completion 2029-05-21 (Estimated)

PRIMARY OUTCOMES:
Best Response | 6 weeks
  The primary objective of the study is to assess the efficacy of early upfront emapalumab on hematologic recovery within 6 weeks of starting therapy after a new diagnosis of Aplastic Anemia. Response will be determined by blood count.

CONTACTS AND LOCATIONS:
Overall Officials: Andromachi Scaradavou, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Cincinnati Children's Hospital Medical Center (Data collection only), Cincinnati, Ohio
  - Children's Hospital of Philadelphia (Data Collection AND Specimen Analysis), Philadelphia, Pennsylvania
  - Virginia Commonwealth University (Data Collection Only ), Richmond, Virginia
  - Children's Hospital of Wisconsin (Data Collection Only), Milwaukee, Wisconsin
  - Medical College of Wisconsin (Data Collection AND Data Analysis), Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org